CLINICAL TRIAL: NCT01397214
Title: A Randomized, Open-label, Single-dose, Cross-over Study to Investigate Safety and Pharmacokinetics of Megace F and Megace OS Under Fasting and Fed Conditions in Healthy Male Volunteers
Brief Title: Pharmacokinetics of Megace F and Megace OS Under Fasting and Fed Conditions in Healthy Male Volunteers
Acronym: MGF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MGF-BR-CT-101
Record Dates: First submitted 2011-07-15; First posted 2011-07-19 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Cachexia; Anorexia
MeSH Terms: conditions — Cachexia; Anorexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Megace F (Experimental): Megace F oral suspension
  Interventions: Drug: Megace F
- Megace OS (Active Comparator): Megace acetate oral suspension
  Interventions: Drug: Megace OS

INTERVENTIONS:
Drug: Megace F — Megace F oral suspension
  Arms: Megace F
Drug: Megace OS — Megace oral suspension
  Arms: Megace OS

SUMMARY:
Phase I study of Megace F will be conducted to investigate pharmacokinetics and safety compared to Megace OS.

Phase I study divided into 3 parts written as belows.

Part 1 Megace F in fasting volunteers vs Megace F in fed volunteers Part 2 Megace F vs Megace OS in fed volunteers Part 3 Megace F vs Megace OS in fasting volunteers

ELIGIBILITY:
Inclusion Criteria:

age: 20-55 years body weight: greater than 50kg written informed consent

Exclusion Criteria:

known allergy to Megesterol acute or chronic diseases which could affect drug absorption or metabolism positive drug or alcohol screening smokers of 10 or more cigarettes per day 3 month ago participation in a clinical trial during the last 3 months prior to the start of the study

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
AUC | 0, 1, 2,3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 hrs

SECONDARY OUTCOMES:
Tmax | 0, 1, 2,3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 hrs
t1/2 | 0, 1, 2,3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, Dr., Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea